CLINICAL TRIAL: NCT03496818
Title: Effect of Small Bowel Crohn's Disease on Chylomicron Secretion After Ingestion of a Fatty Meal
Brief Title: Effect of SB CD on Chylomicron
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201712103
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's Disease: Participants age 18-80 years old, diagnosed with Crohn's disease with active disease based on MR enterography or CT enterography confirmed within the prior 90 days.
- Healthy controls: Participants age 18-80 years old, with no diagnosis of inflammatory bowel disease.

SUMMARY:
It is often suggested that lymphatic vessels are ineffective in transporting cargo in Crohn's disease. Our own work on surgically resected tissue supports this concept (1), but the concept has not been directly tested. Chylomicrons are packaged lipids from the diet with an obligatory absorption route through the lymphatic vasculature to reach host plasma. This protocol takes an approach to directly quantify chylomicron secretion using a fatty meal that incorporates stable isotopic tracers for trioleate and cholesterol in the meal. We will collect baseline plasma and then plasma every 30 minutes for 6 hours to chart the kinetic and magnitude of chylomicron secretion and transport in all subjects using mass spectrometry analysis. We will characterize a wide variety of parameters on the chylomicrons as well using ELISA. Infusions i.v. of stable isotope labeled triglyceride and glycerol will allow us to consider whether there are changes in VLDL metabolism that could account for differences in chylomicron handling once the chylomicrons are secreted into plasma. Collection and analysis of breath samples will also be carried to normalize against possible incomplete lipid absorption in some subjects.

DETAILED DESCRIPTION:
Background:

B1 Prior Literature and Studies Crohn's disease (CD) is characterized by spontaneous, chronic relapsing and remitting inflammation of the gastrointestinal tract. The underlying etiology of the disease is unknown but it likely develops secondary to an environmental stimulus in a genetically predisposed person that results in a dysregulated immune response to the intestinal microbiome. Considerable effort has been paid to understanding the role of the intestinal microbiome, the genetic susceptibilities at play, and the immunology behind the condition to tailor treatments aimed at reducing inflammation.

Prior to the advent of current medical therapies a defining characteristic of CD noted by early pathologists evaluating tissue specimen's was a significant alteration of the gastrointestinal lymphatic system with lymphocytic thrombi, aggregates of lymphocytes and granuloma-obstructed lymphatics consistent with chronic lymphangitis (2). Furthermore, early researchers showed that obstructing segments of the regional lymphatics of the small intestine resulted in a segmental intestinal disease similar to CD (3). Immunohistochemical staining has confirmed the presence of lymphangiectasias, lymphocytic perilymphangitis, lymphocyte or granuloma obstructed lymphatics and inflammatory lymphoid follicles in patients with CD (4). Upstream of these obstructed lymphatics the vessels remain distended with lymphocytes (5). More recent studies have shown that lymphatic density is also significantly increased in the ileal and colonic tissue of patients with CD (6). Furthermore, the relationship between intestinal health and lymphatics has been highlighted in studies that found certain types of bacteria and viruses had resulted in a profoundly remodeled mesenteric lymphatic system. Findings included the development of chronic lymphadenopathy and increased permeability, similar to what is seen in CD (7). Given the prominent structural changes that occur to the mesenteric lymphatic system in CD (1), studies are needed to evaluate if lymphatic function is altered as well.

Chylomicrons are cholesterol and triacylglycerol rich lipoproteins synthesized by the small intestine and transported through the lymphatics. Thus, oral uptake of trioleate and cholesterol will lead to incorporation of the tracers into chylomicrons.

Using ELISA and mass spectrometric analysis these labelled chylomicrons can be quantitated in the serum, thus serving as a marker of absorption and transit through the lymphatics. Studies of healthy subjects have utilized this validated means to assess lymphatic uptake and transport. After ingestion, there is a delay of <60 minutes in the appearance of 13C labelled chylomicrons in the serum, with a peak occurring between 180 and 240 minutes. Our protocol is designed to take advantage of the knowledge that other oral tracer studies at Washington University have learned in optimizing such studies, including ongoing studies by Dr. Todd Cade that focuses on chylomicron secretion in pre-diabetic patients. Our study will evaluate patients with significant small bowel CD and compare them to healthy controls using a similar method.

This pilot study would be the first to evaluate the quantitative function of lymphatics in CD. It would provide the basis for further studies evaluating the mesenteric lymphatics and their role in the pathogenesis of CD and as a treatment target.

C Study Objectives

C1 Primary Aim Follow lymphatic vessel transported cargo in Crohn's disease patients with small bowel involvement as a way to assess possible defects in the lymphatic system in patients compared with healthy control subjects.

C2 Secondary Aim Characterize changes in pre- and post-prandial lipid metabolism resulting from Crohn's disease affecting the small bowel.

C3 Tertiary Aim Carry out lipidomic analyses to determine if chylomicrons absorbed from the small bowel carry distinct microbial lipid signatures compared with healthy control subjects (eg., LPS, commendamide (8)).

C4 Quaternary Aim Measure lipid absorption from the intestine using 13CO2 breath analysis.

D Study Design

D1 Overview or Design Summary This study will utilize a 2-group trial design in which 40 participants (20 CD patients and 20 controls) will visit once for this feeding (oral tracer) and infusion study, following an overnight fast.

Participants will be recruited from the Washington University School of Medicine IBD Center, Washington University's Volunteers for Health, the Center for Community Based Research, and IBD clinics affiliated with Washington University in the surrounding St. Louis community.

The principal investigator, collaborating physicians, and study coordinator(s) will be responsible for identifying participants through the use of posters, email, and existing participant databases.

E Study Procedures

E1 Screening for Eligibility IBD Center staff will identify eligible subjects from the patient arm. By phone, each participant will be asked a series of preliminary screening questions to determine immediate expulsion from the study based on exclusion and inclusion criteria. The purpose of the study, and a brief overview of the procedures, time-commitment, and compensation will be discussed over the phone prior to the individual agreeing to participate.

E2 Study Visit

1. 7:00 AM: Subject reports to the Clinical Research Unit at Washington University School of Medicine.

   1. The subject will be asked to skip breakfast and report to the Clinical Research Unit after an overnight fast (> 8 hours) with nothing taken by mouth except water. Subjects will be asked to avoid caffeine and alcohol for at least 24 h before admission for the study visit. The day prior to the study visit, subjects will be provided instructions for a standardized meal for breakfast, lunch, and dinner containing a total of 2,165 calories (46% of total energy from carbohydrates, 40% from fat, and 14% from protein). A liquid formula (Ensure; Ross Laboratories, Columbus, OH) containing 250 kcal (40 g carbohydrates, 6.1 g fat, and 8.8 g protein) to ensure complete filling of hepatic glycogen stores as a snack before bedtime. This snack is included in the total calories stated above.
   2. The participant will have his/her height and weight measured using the electronic weight scale and stadiometer within the Clinical Research Unit. BMI will be calculated from height and weight using the formula: [mass(kg)/[height(meters)2]. Blood pressure will be measured and recorded.
   3. The participant will complete a medical history questionnaire, which includes obtaining a list of current medications. Completion of the questionnaire may occur following the baseline blood draw and meal administration
2. A catheter will be inserted into the other antecubital vein to obtain blood samples.
3. 8 AM: Metabolism Study: Baseline Period: Baseline blood and breath samples to determine background enrichment of isotopes. Then the subject will then consume a liquid test meal prepared by CRU nutrition staff consisting of 27 g Sol Carb, 1032 g Boost Plus, 3.2 g canola oil, 0.2 g lecithin, 5 mg/kg of [1,2, 3, 7, 8-13C8] glyceryl trioleate, and 40 g of water. Participants will be asked to consume the liquid meal within 20 minutes for consistency, with the sides of the container scraped to ensure maximal ingestion. Additionally, 30 minutes after consuming the meal a 75 micromol/kg bolus infusion of (1,1,2,3,3-2H5)glycerol will be initiated to track VLDL catabolism. Blood and breath samples will be collected at 0, 15. 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes post-meal ingestion. Indirect calorimetry will also be administered using the ventilated hood technique for 10 minutes prior to each breath sample collection to determine resting metabolic rate for tracer calculations and measurement of total fatty acid oxidation. Blood samples will be analyzed for tracer enrichment and total concentration of free fatty acids, triglycerides, and cholesterol.
4. 2 pm: Lunch will be served by CRU, prepared by CRU kitchen. End of Study Visit.

ELIGIBILITY:
Inclusion criteria (experimental group):

1. Age 18-80 year's old.
2. Diagnosed with Crohn's disease.
3. Active small bowel Crohn's disease on MR enterography or CT enterography confirmed within the prior 30 days.
4. Inflammatory markers (eg.,. CRP, ESR) elevated above the upper limit of normal.
5. Ability to provide informed consent.

Inclusion criteria (control group):

1. Age 18-80 years old.
2. Ability to provide informed consent.
3. No diagnosis of inflammatory bowel disease.

Inclusion criteria (inflammatory arthritis or skin inflammation group):

1. Age 18-80 years old.
2. Ability to provide informed consent.
3. Taking a biologic targeting TNF (infliximab, adalimumab) for at least 4 weeks.

Exclusion Criteria

1. A history of diabetes mellitus.
2. A history of hyperlipidemia.
3. A history of thyroid dysfunction.
4. A history of hepatic, cardiac, renal or endocrine dysfunction.
5. A history of cancer requiring systemic chemotherapy
6. Prior radiation therapy to pelvis or abdomen
7. Taking medications (current or past 30 days) known to alter plasma lipid levels including statins, corticosteroids (oral, IV or topical), bile acid sequestrants, thyroid drugs, or fibrates.
8. Currently pregnant or trying to become pregnant.
9. History of abdominal or pelvic surgery.
10. Complicated small bowel CD with obstruction, penetrating disease and/or abscess.
11. Recent surgery of any type within the last 30 days that, in the discretion of the principal investigator, might affect the study or pose risk to the subject

Exclusion for control group: all of the above and no recent participation in other studies as a control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Washington University School of Medicine IBD Center, Washington University's Volunteers for Health, the Center for Community Based Research, and IBD clinics affiliated with Washington University in the surrounding St. Louis community.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Chylomicron transport rate and magnitude | 1 day of Enrollment
  % of meal-delivered triglyceride (trioleate) tracer recovered in the chylomicron fraction of plasma over a 6 h time course will be used to quantify chylomicron transport rate and magnitude

SECONDARY OUTCOMES:
Tracer kinetic calculations | 1 day of Enrollment
  Total plasma triglycerides, cholesterol, free fatty acids will be used for tracer kinetic calculations, as well as to calculate metabolic area under the curves
Maturation of the lipoproteins in plasma | 1 day of Enrollment
  Quantification of plasma apoA-1, apoA-IV, apoB48, apoE, apoCII, apoM and the presence of these proteins in chylomicron, VLDL, LDL, and HDL will serve to characterize the maturation of the lipoproteins in plasma over time in CD versus control samples
NMR analysis | 1 day of Enrollment
  NMR analysis will be used to determine the size of various lipoproteins in the plasma over the time course
Chylomicron secretion | 1 day of Enrollment
  Plasma VEGF-C measurement will be used to determine if chylomicron secretion correlates with release of the lymphatic hormone VEGF-C
Lipid uptake and excretion | 1 day of Enrollment
  % of meal-delivered triglyceride tracer recovered in breath samples will be used to measure exogenous lipid uptake and excretion

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States